CLINICAL TRIAL: NCT06508060
Title: A Randomized Controlled Trial Investigating the Efficacy and Safety of a Device That Uses Bimodal Stimulation, Consisting of Auditory and Vibrotactile Stimuli, for the Mitigation of Tinnitus
Brief Title: Bimodal Stimulation Using Auditory and Vibrotactile Stimuli for the Mitigation of Tinnitus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neosensory (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/01/7
Record Dates: First submitted 2024-07-12; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Tinnitus
Keywords: Biomodal stimulation; Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Tones combined with vibrotactile stimulation (Experimental): The experimental group will receive treatment consisting of tones combined with vibrotactile stimulation delivered from a haptic wristband.
  Interventions: Device: Neosensory Wristband
- Tones alone (Other): The control group will receive treatment consisting of tones alone, without the addition of vibrotactile stimulation from a wristband.
  Interventions: Other: Tones only

INTERVENTIONS:
Device: Neosensory Wristband — The Neosensory wristband consists of four vibratory motors built into the strap of the wristband (Figure 1a). The motors are linear resonant actuators (LRAs), vibrating at 175 Hz, capable of rising from 0 to 50% of their intensity within 30 ms. The motor intensity can be controlled with an eight bit resolution, meaning each motor can be controlled at 256 different intensities. At the highest intensity, each motor vibrates at 1.7 GRMS. The motors are separated from one another at a distance of 18.2 mm and 19.2 mm for the small and large wristband sizes, respectively (center-to-center distances).
  The top of the wristband is a module that contains the power button, user setting buttons, a microphone, and a microcontroller. Bluetooth communication is used to create the corresponding vibrations on the wristband. While the study app plays the tones, it also sends a Bluetooth command to the wristband such that the wristband vibrates in the appropriate illusory location.
  Arms: Tones combined with vibrotactile stimulation
Other: Tones only — Tones will be played through an app
  Arms: Tones alone

SUMMARY:
The goal of this clinical trial is to learn if a bimodal stimulation device that combines auditory tones with vibrotactile stimulation to the wrist works to treat moderate to severe tinnitus in adults. It will also learn about the safety of the device. The main questions it aims to answer are:

1. Does a bimodal stimulation device that combines auditory tones with vibrotactile stimulation to the wrist decrease the severity of tinnitus symptoms in adults with moderate to severe tinnitus?
2. What medical problems do participants report when using a bimodal stimulation device that combines auditory tones with vibrotactile stimulation to the wrist?

Researchers will compare a bimodal stimulation device that combines auditory tones with vibrotactile stimulation to the wrist to a control condition in which only auditory tones are used, without the device, to see if the bimodal stimulation device works to treat moderate to severe tinnitus.

Participants will:

1. Use the bimodal stimulation device for 10 minutes every day for a period of 8 weeks
2. Have one-on-one calls with the research team at the beginning and end of the study
3. Complete baseline and final tinnitus functional index assessments to track progress as a result of the intervention.

DETAILED DESCRIPTION:
Our research hypothesis is, randomized tones coupled with a spatial spread of vibrotactile signals on the wrist to deliver bimodal stimulation will decrease the severity of tinnitus symptoms as measured by a clinically significant improvement on the Tinnitus Functional Index questionnaire (TFI). We also hypothesize this treatment will prove to be safe, with minimal or no side effects.

We will recruit adults in the United States who respond to an online advertisement that mentions a study investigating a new tinnitus treatment. A total of 200 participants will be confirmed and randomly assigned to a wristband condition or an audio-only control condition (100 participants per condition).

Each participant will complete ten minutes of treatment daily over the course of the eight-week study. The treatment will include listening to tones and, unless in the control condition, feeling corresponding vibrations on the wrist. In the control condition, participants will listen to tones without additional vibrotactile stimulation from a wristband. Participants will complete the TFI questionnaire at baseline prior to starting treatment with Duo and after 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide and understand informed consent
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Initial Tinnitus Functional Index Score of 42 points or higher indicating mild, moderate, or severe tinnitus
* Subjective tinnitus that is described as tonal or white noise
* Age 22 and over at the time of consent
* Ability to read and understand English
* Tinnitus duration for greater than or equal to 3 months
* Able to provide an audiogram performed by a licensed audiologist within the past 12 months

Exclusion Criteria:

* Individuals who are non-English speaking
* Subjective tinnitus, where pulsatility is the dominant feature (participant reported)
* Objective tinnitus, where the tinnitus is also observed by the examiner
* Commenced usage of hearing aid within the last 90 days
* Meniere's disease
* Hospitalization, or visit to a physician, for a head or neck injury, including whiplash, in the previous 12 months
* TMJ Disorder
* Pregnancy
* Neurological condition that may lead to seizures or loss of consciousness (e.g. epilepsy)
* Severe cognitive impairment based on MMSE (score less than 20)
* Abnormal findings following otoscopy/tympanometry that may be contributing to or causing the tinnitus as assessed by an Audiologist/ENT (participant reported)
* Initiated new prescription medications or medical treatments in the previous 3 months
* Ceased prescription medications or medical treatments in the previous 3 months
* Participant previously diagnosed with psychosis or schizophrenia
* Previous use of Neosensory Duo
* Previous involvement in a clinical investigation for tinnitus or had an experimental/surgical treatment for tinnitus
* Hearing loss of greater than 80 dB HL in any test frequency in the set {2k,3k,4k,6k,8k} Hz or greater than 40 dB HL in the set {250,500,1k} Hz either unilaterally or bilaterally. This information will be obtained from an audiogram performed by a licensed audiologist, that is provided by the candidate.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Functional Index | From the first day of treatment to the final day of treatment at 8 weeks
  The Tinnitus Functional Index (TFI) is a self-report questionnaire that measures the severity and negative effects of tinnitus. It's used to assess how tinnitus affects a person in multiple domains, and can also be used to measure changes in tinnitus related to treatment.

IPD SHARING:
Plan to Share IPD: No
We have no reason to share IPD with other researchers